CLINICAL TRIAL: NCT07288567
Title: A Phase 3 Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of KarXT for the Treatment of Schizophrenia in Adolescents (13 to 17 Years of Age)
Brief Title: A Study to Evaluate the Efficacy and Safety of KarXT for the Treatment of Schizophrenia in Adolescents
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CN012-0020; 2025-523711-11-00 (Other: EU CT number); U1111-1325-9936 (Other: WHO)
Record Dates: First submitted 2025-12-16; First posted 2025-12-17 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KarXT (Experimental)
  Interventions: Drug: KarXT
- Placebo (Placebo Comparator)
  Interventions: Other: KarXT Matching Placebo

INTERVENTIONS:
Drug: KarXT — Specified dose on specified days
  Other Names: BMS-986510
  Arms: KarXT
Other: KarXT Matching Placebo — Specified dose on specified days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of KarXT for treatment of Schizophrenia in adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia as defined by the The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition,Text Revision (DSM-5-TR) criteria, confirmed by the Kiddie Schedule for Affective Disorders and Schizophrenia-Present and Lifetime version (K-SADS-PL) and experiencing symptoms of psychosis at screening (Visit 1).
* PANSS total score of at least 70 at screening (Visit 1) and randomization (Visit 2).
* Participant has a CGI-S score of ≥ 4 at screening (Visit 1) and randomization (Visit 2).

Exclusion Criteria:

* Any primary DSM-5-TR disorder other than schizophrenia within 12 months before screening.
* History or presence of clinically significant cardiovascular, pulmonary, hepatic impairment, renal, hematologic, GI, endocrine, immunologic, dermatologic, neurologic, or oncologic disease or any other condition that, in the opinion of the investigator, would jeopardize the safety of the participant or the validity of the study results.
* All grades of hepatic impairment (mild [Child-Pugh Class A], moderate [Child-Pugh Class B], and severe [Child-Pugh Class C]). Participants with known intellectual disability defined as an IQ less than 70; or, either clinical evidence or known social or school history indicative of intellectual disability.
* Any neurological disorder, except for Tourette's Syndrome.
* Participants who have either a systolic blood pressure (sBP) or diastolic blood pressure (dBP) meeting criteria for stage 2 HTN, regardless of the presence or absence of symptoms.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 166 (Estimated)
Dates: Start 2026-01-29 (Actual); Primary Completion 2029-12-18 (Estimated); Study Completion 2029-12-18 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score | Week 5

SECONDARY OUTCOMES:
Change From Baseline in Clinical Global Impression-Severity (CGI-S) Score | Week 5
Change From Baseline in PANSS Positive Subscale Score | Week 5
Change From Baseline in PANSS Negative Subscale Score | Week 5
Change From Baseline in PANSS Marder Negative Factor Score | Week 5
Number of Participants With PANSS Response | Week 5
  PANSS response will be determined by ≥ 30% reduction in PANSS total score.
Change From Baseline in Clinical Global Impression - Improvement (CGI-I) Score | Week 5
Change From Baseline in Children's Global Assessment Scale (CGAS)) Score | Week 5

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (43):
- United States (20):
  - Local Institution - 0077, Anaheim, California
  - Local Institution - 0058, Chino, California
  - Local Institution - 0089, San Francisco, California
  - Local Institution - 0032, Orlando, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Local Institution - 0106, Lawrenceville, Georgia
  - Local Institution - 0039, Stone Mountain, Georgia
  - Local Institution - 0044, Chicago, Illinois
  - Local Institution - 0107, Evanston, Illinois
  - Local Institution - 0076, Boston, Massachusetts
  - Local Institution - 0100, Brookline, Massachusetts
  - Local Institution - 0059, Worcester, Massachusetts
  - Local Institution - 0049, Highland Park, Michigan
  - Local Institution - 0061, Great Neck, New York
  - Local Institution - 0051, Cincinnati, Ohio
  - Local Institution - 0099, Philadelphia, Pennsylvania
  - Local Institution - 0046, Garland, Texas
  - Local Institution - 0090, McAllen, Texas
  - Local Institution - 0066, Spring, Texas
  - Local Institution - 0050, Richmond, Virginia
- Argentina (5):
  - Local Institution - 0084, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Local Institution - 0085, La Plata, Buenos Aires
  - Local Institution - 0036, Buenos Aires
  - Local Institution - 0035, Córdoba
  - Local Institution - 0102, Santiago del Estero
- Colombia (3):
  - Local Institution - 0009, Pereira, Risaralda Department
  - Local Institution - 0001, Barranquilla
  - Local Institution - 0020, Bogotá
- Japan (7):
  - Local Institution - 0075, Chikugo-Shi, Fukuoka
  - Local Institution - 0073, Sapporo, Hokkaido
  - Local Institution - 0025, Zentsujichó, Kagawa-ken
  - Local Institution - 0062, Miyakonojō, Miyazaki
  - Local Institution - 0086, Bunkyo-ku, Tokyo
  - Local Institution - 0056, Ōta-ku, Tokyo
  - Local Institution - 0063, Yokohama, Kanagawa
- Romania (8):
  - Local Institution - 0029, Bucharest, București
  - Local Institution - 0031, Brasov
  - Local Institution - 0040, Bucharest
  - Local Institution - 0042, Bucharest
  - Local Institution - 0008, Iași
  - Local Institution - 0030, Sibiu
  - Local Institution - 0005, Timișoara
  - Local Institution - 0038, Timișoara

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT07288567.html